CLINICAL TRIAL: NCT06076226
Title: The First Affiliated Hospital, Zhejiang University School of Medicine
Brief Title: A Retrospective Study on the Relationship Between Donor Leukocyte Telomere Length and Prognosis of Acute Leukemia Patients Treated With Allogeneic Hematopoietic Stem Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, The President of the First Affiliated Hospital, Zhejiang University School of Medicine, Zhejiang University
Other Study IDs: Telo-2015-HSCT
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Donors aged 40 years or older
  Interventions: Other: No intervention, observation study
- Donors aged < 40
  Interventions: Other: No intervention, observation study

INTERVENTIONS:
Other: No intervention, observation study — No intervention, observation study

SUMMARY:
This post hoc analysis included patients with acute leukemia who underwent allo-HSCT at the First Affiliated Hospital of Zhejiang University School of Medicine and Ruijin Hospital Shanghai Jiaotong University School of Medicine. Patients and their donors were assessed for eligibility to join this study. The inclusion criteria were: (1) age ≥ 5 years; (2) diagnosis of acute leukemia including acute myeloid leukemia, acute lymphocytic leukemia, and mixed phenotype acute leukemia; (3) patients attained complete remission (CR) and achieved full engraftment with 100% donor chimerism following allo-HSCT; (4) telomere testing was conducted on peripheral leukocytes of donors before granulocyte colony-stimulating factor (G-CSF) mobilization, and the results were obtained. Written informed consent was obtained from all included patients and their donors, and the study was conducted in compliance with the Declaration of Helsinki. Ethical approval was approved by the ethics review committee of the First Affiliated Hospital of Zhejiang University School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years
* First allo-HSCT from matched related, unrelated, or haploidentical donors
* Achievement of complete remission after allo-HSCT
* Donor blood sample collection before granulocyte colony-stimulating factor mobilization

Exclusion Criteria

* Non-acute leukemia diagnoses, including acute myeloid leukemia, acute lymphocytic leukemia, and mixed phenotype acute leukemia
* Failure to achieve engraftment with full donor chimerism after allo-HSCT
* Inability to extract DNA for telomere length analysis.

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study aims to investigate the influence of donor blood telomere length on recipients' clinical outcomes post-allogeneic hematopoietic stem cell transplant.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of transplantuntil the date of death from any cause, assessed up to 60 months.
  The duration from transplant until death resulted from any cause.

SECONDARY OUTCOMES:
Relapse-free survival | From date of transplant until the date of relapse or death from any cause, assessed up to 60 months.
  The time from transplant until death or relapse.
Cumulative incidence of relapse | From date of transplant until the date of relapse, assessed up to 60 months.
  The time interval between the transplant and the occurrence of relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical research ethics committee of the first affiliated hospital, college of medicine, zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No